CLINICAL TRIAL: NCT03668678
Title: iGrow Readers Nutrition and Physical Activity Curriculum Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Dakota State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jessica Meendering, Associate Professor, South Dakota State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1408008; 2011-67002-30202 (Other: USDA National Institute of Food and Agriculture)
Record Dates: First submitted 2018-09-07; First posted 2018-09-12 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Pediatric Obesity; Knowledge, Attitudes, Practice; Physical Activity; Diet Modification
Keywords: Obesity; Physical Activity; Nutrition; Curriculum; Preschool; Literacy
MeSH Terms: conditions — Pediatric Obesity; Behavior; Motor Activity; Obesity; Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iGrow Readers Curriculum (Experimental): The iGrow Readers nutrition and physical activity curriculum was implemented in early-childhood classrooms assigned to the IGrow Readers intervention group.
  Interventions: Other: iGrow Readers Curriculum
- Standard Curriculum (No Intervention): The standard curriculum was provided within early-childhood classrooms assigned to the control group.

INTERVENTIONS:
Other: iGrow Readers Curriculum — As part of the iGrow Readers curriculum, the primary teacher first reads a book as a group with a specific health behavior theme. Then, children participate in nutrition and physical activities that relate and reinforce the lessons learned in the book. Informational newsletters highlighting healthy behaviors from the stories' themes are provided to parents. All implementation strategies are reinforced by research to promote positive choices in young children's health behaviors through the use of literature and language strategies and modeling of others in the children's microsystems.
  Arms: iGrow Readers Curriculum

SUMMARY:
The objective of this study was to determine the efficacy of the iGrow Readers curriculum in changing diet and physical activity knowledge among preschool-aged children. The secondary objective of this study was to better understand the relationship between diet and physical activity related outcome variables in preschool aged children and their primary caregivers.

DETAILED DESCRIPTION:
The objective of this study was to determine the efficacy of the iGrow Readers curriculum in changing diet and physical activity knowledge among preschool-aged children. The secondary objective of this study was to better understand the relationship between diet and physical activity related outcome variables in preschool aged children and their primary caregivers.

iGrow Readers was created to support literacy development among preschoolers, while promoting nutrition and physical activity messages. This program utilizes the social cognitive theory because it focuses on different environments influencing individual's behaviors and knowledge acquisitions, primarily through observing others within the context of social interactions and experiences. Developmentally appropriate preschool-aged children books, including relevant Native American books, facilitate the themes of healthy physical activity and nutrition practices. The program, a 6-8-week educational curriculum, helps young children understand the benefits of making healthy decisions involving nutrition and physical activity.

ELIGIBILITY:
Inclusion Criteria:

3-5 year old children attending a participating early childhood care facility. All early childhood care facilities had at least two classrooms available. All children provided assent and their participating guardian provided consent.

Exclusion Criteria:

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 568 (Actual)
Dates: Start 2014-08-14 (Actual); Primary Completion 2016-08-13 (Actual); Study Completion 2016-08-13 (Actual)

PRIMARY OUTCOMES:
Change in Nutrition and Physical Activity Knowledge | Data was collected prior to delivering the curriculum (pre-intervention), from 6-13 weeks after the intervention (post-intervention), and 24-33 weeks following the completion of the intervention (follow-up).
  The Child Nutrition and Physical Activity Survey Tool was used for assessment of nutrition and physical activity knowledge in children.

SECONDARY OUTCOMES:
Change in Height | Data was collected prior to delivering the curriculum (pre-intervention), from 6-13 weeks after the intervention (post-intervention), and 24-33 weeks following the completion of the intervention (follow-up)
  Height was measured in cm via shorrboard.
Change in Weight | Data was collected prior to delivering the curriculum (pre-intervention), from 6-13 weeks after the intervention (post-intervention), and 24-33 weeks following the completion of the intervention (follow-up)
  Weight was measured in kg on an electronic scale.
Change in Body Composition - Lean mass and fat mass | Data was collected prior to delivering the curriculum (pre-intervention), from 6-13 weeks after the intervention (post-intervention), and 24-33 weeks following the completion of the intervention (follow-up)
  Lean mass and fat mass were measured with bio-electrical impedance analysis in children, their guardian, and their teacher.
Change in Body Mass Index | Data was collected prior to delivering the curriculum (pre-intervention), from 6-13 weeks after the intervention (post-intervention), and 24-33 weeks following the completion of the intervention (follow-up)
  Body Mass Index (kg/m^2) was calculated in adults and Body Mass Index Percentile was calculated in children.
Teacher Perceptions of the Curriculum | up to 33 weeks
  The Teacher Feedback Questionnaire was used to evaluate teacher perceptions, ideas, and events related to iGrow Readers. The questionnaire consisted of 26 questions that asked teachers about the changes they may have noticed in their children and themselves, and if they modeled nutrition-based changes for their children after the program's implementation. In addition, teachers were asked to rate the children's responsiveness to the program, if they planned to spend more time on nutrition and PA education in the classroom, and what components of the program the teachers and children enjoyed the most.
Change in Physical Activity | Data was collected prior to delivering the curriculum (pre-intervention), from 6-13 weeks after the intervention (post-intervention), and 24-33 weeks following the completion of the intervention (follow-up)
  Accelerometers were used for assessment of physical activity in children, their guardian, and their teacher.
Change in Sedentary Behavior | Data was collected prior to delivering the curriculum (pre-intervention), from 6-13 weeks after the intervention (post-intervention), and 24-33 weeks following the completion of the intervention (follow-up)
  Accelerometers were used for assessment of sedentary behavior in children, their guardian, and their teacher.
Change in Diet | Data was collected prior to delivering the curriculum (pre-intervention), from 6-13 weeks after the intervention (post-intervention), and 24-33 weeks following the completion of the intervention (follow-up)
  The Harvard Service Food Frequency Questionnaire (HSFFQ) was used to assess dietary behaviors and was completed by teachers and guardians. Teachers provided responses about themselves and the guardians provided responses about themselves and on behalf of their child. The questionnaire lists 87 different food items for adults (86 for children) and ask the number of times the food was consumed during the past 4 weeks. Each food item has a response scale of 0 to 8 (0 = "Never"; 1 = "1-3 times/month"; 2 = "1 time/week"; 3 = "2-4 times/week"; 4 = "5-6 times/week"; 5 = "1 time/day"; 6 = "2-3 times/day"; 7 = "4-5 times/day"; and 8 = "more than 6 times/day").
Home Environment - Nutrition and Physical Activity | up to 33 weeks
  The home environment was assessed via the comprehensive home environment survey.
Caregiver physical activity practices | up to 33 weeks
  Caregiver physical activity practices were assessed via the parent report version of the Activity Support Scale for Multiple Groups (ACTS-MG). The ACTS-MG measures parental support for children's physical activity and includes the following sub-scales: modeling, logistical support, and restricting access to screen-based activities. Each of the 20 items on the questionnaire has a response scale of 1 (strongly disagree) to 4 (strongly agree). The overall score is a mean score across all questions and subscale scores are mean scores of the questions within the subscale. The higher the score, the greater the parental support for physical activity of the child.
Parenting Style | up to 33 weeks
  The parenting dimensions inventory was used to assess parenting style in guardians.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Meendering, PhD, Principal Investigator — South Dakota State University

IPD SHARING:
Plan to Share IPD: Undecided
The research team has not determined if the individual participant data will be made available to other researchers at this time as we are still actively publishing from this dataset.